CLINICAL TRIAL: NCT04095507
Title: Efficacy and Efficiency of Uterocervical Angle for Prediction of Labor Timing in Patients With Preterm Premature Rupture of the Membranes: a Prospective Cohort Study
Brief Title: Uterocervical Angle in Patients With Preterm Premature Rupture of the Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nefise Nazlı YENIGUL (Other)
Responsible Party: Sponsor-Investigator, Nefise Nazlı YENIGUL, Principal Investigator, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10987
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uterocervical angle (Other): uterocervical angle is the angle between lower segment of uterus and cervix
  Interventions: Diagnostic Test: uterocervical angle

INTERVENTIONS:
Diagnostic Test: uterocervical angle — uterocervical angle is the angle between lower segment of uterus and cervix

SUMMARY:
To evaluate the performance of uterocervical angle (UCA) in the prediction of labor timing in patients with preterm premature rupture of the membranes

ELIGIBILITY:
Inclusion Criteria:

* no previous systemic illnesses
* Preterm Premature Rupture of the Membranes

Exclusion Criteria:

* abnormal Pap smear
* previous cesarean section
* history of dilatation and curettage (D&C)
* history of loop electrosurgical excision procedure (LEEP) and cervical conization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
prediction of birth timing by uterocervical angle in patients with Preterm Premature Rupture of the Membranes | 7 month]
  During the study period, women were enrolled and uterocervical angle were measured in the first evaluations of polyhydramnios patients in policlinics. Routine pregnancy follow-up was done by our team and weeks of delivery and maternal-fetal outcomes were noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanliurfa Traning and Research Hospital, Sanliurfa, Turkey (Türkiye)